CLINICAL TRIAL: NCT05760157
Title: To Establish a Multimodal Dynamic Risk Assessment System of Heart Failure in Patients With Myocardial Infarction Based on Coronary Microcirculation.
Brief Title: Mulltimodal Dynamic Risk Assessment Systems of Heart Failure in Patients With Myocardial Infarction.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jian Liu (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Anzhen Hospital (Other); Navy General Hospital, Beijing (Other); Beijing Luhe Hospital (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor-Investigator, Jian Liu, Medical Doctor, Chief physician, Professor of Medicine of PUHSC, Doctorial supervisor of PUHSC, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: RDGS2022-08
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure; Acute Myocardial Infarction
Keywords: acute myocardial infarction; heart failure; dysfunction of coronary microcirculation; risk assessment
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling cohort: The first 425(425/567,75%) patients with acute ST-segment elevation myocardial infarction were used to establish a heart failure risk prediction model.
  Interventions: Other: Possible risk factors of heart failure
- Validation cohort: The latter 142(142/567,25%) patients with acute ST-segment elevation myocardial infarction were used to further validate the validity and predictive power of the risk model
  Interventions: Other: Possible risk factors of heart failure

INTERVENTIONS:
Other: Possible risk factors of heart failure — Demographic data, previous medical history data, physical examination, ECG examination, blood routine, blood biochemistry, the peak value of myocardial injury markers, serum markers of heart failure, high-sensitivity C-reactive protein Coronary angiography, interventional treatment, microcirculation resistance index caIMR calculation based on coronary angiography Doppler echocardiography, medication during hospitalization, NYHA cardiac function grading before discharge, and 6-minute walk test before discharge.

SUMMARY:
This study aims to explore the heart failure risk model based on the dynamic data of patients with different outcome nodes after myocardial infarction to correct the heart failure risk of patients timely.

DETAILED DESCRIPTION:
Heart failure (HF) is the most common complication of acute myocardial infarction (AMI), which seriously affects the prognosis and quality of life of patients. After successful revascularization, the risk of heart failure in patients with acute myocardial infarction is closely related to the state of coronary microcirculation, and the risk of heart failure also changes dynamically with the prognosis of patients. However, current heart failure prediction models only include routine baseline variables to assess short-and long-term risk and lack newly explored new risk factors for heart failure-coronary microcirculation function, there are static, single defects. Therefore, this study is intended to be based on patients with acute ST-segment elevation myocardial infarction who had an infarct artery in the anterior descending artery and underwent emergency percutaneous coronary intervention to open the culprit lesion within 12 hours, according to the multi-dimensional data of clinical epidemiology, serology, radiology, and microcirculation resistance index based on coronary angiography during hospitalization and 6 and 12 months after discharge, respectively, to construct a multimodal dynamic predictive model for heart failure risk at 0-24 months, 6-24 months, and 12-24 months after acute myocardial infarction, to explore the heart failure risk model based on the dynamic data of different outcome nodes of patients after myocardial infarction, and to achieve the goal of timely correction of heart failure risk of patients, which is multi-linear, dynamic and practical, to provide a stage-by-stage reference for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including threshold), gender unlimited
2. acute ST-segment elevation myocardial infarction was diagnosed, and the following two criteria were met: A) ischemic chest pain lasting ≥30 min；B) ECG indicating ST-segment elevation ≥0.1 mV in two or more limb leads and/or ≥0.2 mV in two or more adjacent chest leads
3. Coronary angiography confirmed that the culprit's vessel was located in the anterior descending branch, and the proximal and middle segments of the anterior descending branch were occluded (TIMI blood flow 0 or 1), Or TIMI blood flow grade 2 with obvious thrombus (TIMI thrombus score ≥ 2 points, which is determined after the guide wire passes and restores the forward blood flow. The TIMI thrombus score is determined as follows: 0 point: no thrombus is determined；1 point: blurred thrombus image is visible；2 point: clear thrombus image, but the length of the thrombus image is less than 1/2 vessel diameter；3 point: clear thrombus image, the length of the thrombus image is 1/2~2 times the vessel diameter；4 point: clear thrombus image, the thrombus image is more than 2 times the vessel diameter；5 points : complete occlusion of blood vessels)

4：Emergency PCI revascularization was completed within 12 hours after the occurrence of myocardial infarction. Postoperative angiography confirmed that residual stenosis was less than 50%.

5: Sign the informed consent form voluntarily

Exclusion Criteria:

1. Severe heart failure at discharge (NYHA III/IV, EF<30%)；Or patients with severe hemodynamic instability and cardiogenic shock, defined as systolic blood pressure<90 mmHg, and/or cardiac index<2.2 L/min/m2 during continuous (>30 minutes) attacks, identified as secondary cardiac insufficiency, and/or requiring extraintestinal muscle strength or vasoconstrictor or mechanical support to maintain blood pressure and cardiac index above these specified levels.
2. patients undergoing coronary artery bypass grafting
3. Patients with mechanical complications after myocardial infarction
4. prolonged or invasive cardiopulmonary resuscitation
5. Patients with acute pericarditis, infective endocarditis, severe valvular heart disease and cardiomyopathy
6. Serious liver and kidney failure and other diseases, mental disorders or cognitive disorders
7. The expected survival of tumor patients is less than 2 years
8. patients who are participating in other interventional clinical trials
9. Those who refuse to participate or are clearly unable to complete the follow-up according to the established time point.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2023 to December 2023, the patients with acute ST-segment elevation myocardial infarction whose anterior descending branch is the infarcted artery were selected consecutively by the People's Hospital of Peking University, the Third Hospital of Peking University, Anzhen Hospital affiliated to Capital Medical University, the Sixth Medical Center of the General Hospital of the People's Liberation Army, Beijing Luhe Hospital, and Beijing Chaoyang Hospital
Sampling Method: Non-Probability Sample
Enrollment: 567 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of death or re-admission due to heart failure or aggravation of heart failure symptoms. | Within 24 months after discharge
  Readmission due to heart failure was defined as admission with a primary diagnosis of heart failure presenting as a new or worsening heart failure symptom or sign accompanied by elevated natriuretic peptide levels or objective evidence of imaging suggestive of pulmonary systemic congestion; He was treated for heart failure during his hospital stay. Heart failure symptoms aggravate refers to aggravate to New York cardiac function class (NYHA) III/IV

SECONDARY OUTCOMES:
Changes in left ventricular ejection fraction | Within 24 months after discharge
  The difference in left ventricular ejection fraction during follow-up
The change of BNP/NT-pro-BNP. | Within 24 months after discharge
  The difference in BNP/NT-pro-BNP during follow-up
Changes in 6-minute walking experiment. | Within 24 months after discharge
  Distance difference of 6-minute walking test during follow-up
Changes in patients' subjective quality of life score | Within 24 months after discharge
  The difference in quality of life scores during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jian Liu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Jian Liu, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share personal data.

REFERENCES:
- [Background] Ezekowitz JA, Kaul P, Bakal JA, Armstrong PW, Welsh RC, McAlister FA. Declining in-hospital mortality and increasing heart failure incidence in elderly patients with first myocardial infarction. J Am Coll Cardiol. 2009 Jan 6;53(1):13-20. doi: 10.1016/j.jacc.2008.08.067. PMID 19118718
- [Background] Bozkurt B, Coats AJ, Tsutsui H, Abdelhamid M, Adamopoulos S, Albert N, Anker SD, Atherton J, Bohm M, Butler J, Drazner MH, Felker GM, Filippatos G, Fonarow GC, Fiuzat M, Gomez-Mesa JE, Heidenreich P, Imamura T, Januzzi J, Jankowska EA, Khazanie P, Kinugawa K, Lam CSP, Matsue Y, Metra M, Ohtani T, Francesco Piepoli M, Ponikowski P, Rosano GMC, Sakata Y, SeferoviC P, Starling RC, Teerlink JR, Vardeny O, Yamamoto K, Yancy C, Zhang J, Zieroth S. Universal Definition and Classification of Heart Failure: A Report of the Heart Failure Society of America, Heart Failure Association of the European Society of Cardiology, Japanese Heart Failure Society and Writing Committee of the Universal Definition of Heart Failure. J Card Fail. 2021 Apr;27(4):387-413. doi: 10.1016/j.cardfail.2021.01.022. Epub 2021 Mar 1. PMID 33663906
- [Background] Shah RV, Holmes D, Anderson M, Wang TY, Kontos MC, Wiviott SD, Scirica BM. Risk of heart failure complication during hospitalization for acute myocardial infarction in a contemporary population: insights from the National Cardiovascular Data ACTION Registry. Circ Heart Fail. 2012 Nov;5(6):693-702. doi: 10.1161/CIRCHEARTFAILURE.112.968180. Epub 2012 Oct 9. PMID 23051950
- [Background] Ali AS, Rybicki BA, Alam M, Wulbrecht N, Richer-Cornish K, Khaja F, Sabbah HN, Goldstein S. Clinical predictors of heart failure in patients with first acute myocardial infarction. Am Heart J. 1999 Dec;138(6 Pt 1):1133-9. doi: 10.1016/s0002-8703(99)70080-3. PMID 10577445
- [Background] Granger CB, Goldberg RJ, Dabbous O, Pieper KS, Eagle KA, Cannon CP, Van De Werf F, Avezum A, Goodman SG, Flather MD, Fox KA; Global Registry of Acute Coronary Events Investigators. Predictors of hospital mortality in the global registry of acute coronary events. Arch Intern Med. 2003 Oct 27;163(19):2345-53. doi: 10.1001/archinte.163.19.2345. PMID 14581255
- [Background] Bahit MC, Kochar A, Granger CB. Post-Myocardial Infarction Heart Failure. JACC Heart Fail. 2018 Mar;6(3):179-186. doi: 10.1016/j.jchf.2017.09.015. PMID 29496021
- [Background] Zheng H, Foo LL, Tan HC, Richards AM, Chan SP, Lee CH, Low AFH, Hausenloy DJ, Tan JWC, Sahlen AO, Ho HH, Chai SC, Tong KL, Tan DSY, Yeo KK, Chua TSJ, Lam CSP, Chan MY. Sex Differences in 1-Year Rehospitalization for Heart Failure and Myocardial Infarction After Primary Percutaneous Coronary Intervention. Am J Cardiol. 2019 Jun 15;123(12):1935-1940. doi: 10.1016/j.amjcard.2019.03.021. Epub 2019 Mar 19. PMID 30979413
- [Background] Camici PG, d'Amati G, Rimoldi O. Coronary microvascular dysfunction: mechanisms and functional assessment. Nat Rev Cardiol. 2015 Jan;12(1):48-62. doi: 10.1038/nrcardio.2014.160. Epub 2014 Oct 14. PMID 25311229
- [Background] Rush CJ, Berry C, Oldroyd KG, Rocchiccioli JP, Lindsay MM, Touyz RM, Murphy CL, Ford TJ, Sidik N, McEntegart MB, Lang NN, Jhund PS, Campbell RT, McMurray JJV, Petrie MC. Prevalence of Coronary Artery Disease and Coronary Microvascular Dysfunction in Patients With Heart Failure With Preserved Ejection Fraction. JAMA Cardiol. 2021 Oct 1;6(10):1130-1143. doi: 10.1001/jamacardio.2021.1825. PMID 34160566
- [Background] Xie F, Qian L, Goldsweig A, Xu D, Porter TR. Event-Free Survival Following Successful Percutaneous Intervention in Acute Myocardial Infarction Depends on Microvascular Perfusion. Circ Cardiovasc Imaging. 2020 Jun;13(6):e010091. doi: 10.1161/CIRCIMAGING.119.010091. Epub 2020 Jun 12. PMID 32527159
- [Background] Gaibazzi N, Reverberi C, Lorenzoni V, Molinaro S, Porter TR. Prognostic value of high-dose dipyridamole stress myocardial contrast perfusion echocardiography. Circulation. 2012 Sep 4;126(10):1217-24. doi: 10.1161/CIRCULATIONAHA.112.110031. Epub 2012 Aug 7. PMID 22872314
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Tebaldi M, Biscaglia S, Di Girolamo D, Erriquez A, Penzo C, Tumscitz C, Campo G. Angio-Based Index of Microcirculatory Resistance for the Assessment of the Coronary Resistance: A Proof of Concept Study. J Interv Cardiol. 2020 Oct 25;2020:8887369. doi: 10.1155/2020/8887369. eCollection 2020. PMID 33162844
- [Background] De Maria GL, Scarsini R, Shanmuganathan M, Kotronias RA, Terentes-Printzios D, Borlotti A, Langrish JP, Lucking AJ, Choudhury RP, Kharbanda R, Ferreira VM; Oxford Acute Myocardial Infarction (OXAMI) Study Investigators; Channon KM, Garcia-Garcia HM, Banning AP. Angiography-derived index of microcirculatory resistance as a novel, pressure-wire-free tool to assess coronary microcirculation in ST elevation myocardial infarction. Int J Cardiovasc Imaging. 2020 Aug;36(8):1395-1406. doi: 10.1007/s10554-020-01831-7. Epub 2020 May 14. PMID 32409977
- [Background] Choi KH, Dai N, Li Y, Kim J, Shin D, Lee SH, Joh HS, Kim HK, Jeon KH, Ha SJ, Kim SM, Jang MJ, Park TK, Yang JH, Song YB, Hahn JY, Doh JH, Shin ES, Choi SH, Gwon HC, Lee JM. Functional Coronary Angiography-Derived Index of Microcirculatory Resistance in Patients With ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2021 Aug 9;14(15):1670-1684. doi: 10.1016/j.jcin.2021.05.027. PMID 34353599
- [Background] Lazzarini V, Mentz RJ, Fiuzat M, Metra M, O'Connor CM. Heart failure in elderly patients: distinctive features and unresolved issues. Eur J Heart Fail. 2013 Jul;15(7):717-23. doi: 10.1093/eurjhf/hft028. Epub 2013 Feb 20. PMID 23429975
- [Background] Bulluck H, Zheng H, Chan MY, Foin N, Foo DC, Lee CW, Lim ST, Sahlen A, Tan HC, Tan JW, Tong KL, Wong AS, Wong PE, Yeo KK, Foo LL, Chua TS, Koh TH, Hausenloy DJ. Independent Predictors of Cardiac Mortality and Hospitalization for Heart Failure in a Multi-Ethnic Asian ST-segment Elevation Myocardial Infarction Population Treated by Primary Percutaneous Coronary Intervention. Sci Rep. 2019 Jul 11;9(1):10072. doi: 10.1038/s41598-019-46486-0. PMID 31296912
- [Background] Schnabel RB, Rienstra M, Sullivan LM, Sun JX, Moser CB, Levy D, Pencina MJ, Fontes JD, Magnani JW, McManus DD, Lubitz SA, Tadros TM, Wang TJ, Ellinor PT, Vasan RS, Benjamin EJ. Risk assessment for incident heart failure in individuals with atrial fibrillation. Eur J Heart Fail. 2013 Aug;15(8):843-9. doi: 10.1093/eurjhf/hft041. Epub 2013 Apr 17. PMID 23594831
- [Background] Wong YW, Thomas L, Sun JL, McMurray JJ, Krum H, Hernandez AF, Rutten GE, Leiter LA, Standl E, Haffner SM, Mazzone T, Martinez FA, Tognoni G, Giles T, Califf RM. Predictors of incident heart failure hospitalizations among patients with impaired glucose tolerance: insight from the Nateglinide And Valsartan in Impaired Glucose Tolerance Outcomes Research study. Circ Heart Fail. 2013 Mar;6(2):203-10. doi: 10.1161/CIRCHEARTFAILURE.112.000086. Epub 2013 Feb 6. PMID 23388113
- [Background] Agarwal SK, Chambless LE, Ballantyne CM, Astor B, Bertoni AG, Chang PP, Folsom AR, He M, Hoogeveen RC, Ni H, Quibrera PM, Rosamond WD, Russell SD, Shahar E, Heiss G. Prediction of incident heart failure in general practice: the Atherosclerosis Risk in Communities (ARIC) Study. Circ Heart Fail. 2012 Jul 1;5(4):422-9. doi: 10.1161/CIRCHEARTFAILURE.111.964841. Epub 2012 May 15. PMID 22589298
- [Background] Sulo G, Igland J, Vollset SE, Nygard O, Ebbing M, Sulo E, Egeland GM, Tell GS. Heart Failure Complicating Acute Myocardial Infarction; Burden and Timing of Occurrence: A Nation-wide Analysis Including 86 771 Patients From the Cardiovascular Disease in Norway (CVDNOR) Project. J Am Heart Assoc. 2016 Jan 7;5(1):e002667. doi: 10.1161/JAHA.115.002667. PMID 26744379
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Yoon GS, Ahn SG, Woo SI, Yoon MH, Lee MJ, Choi SH, Seo JY, Kwon SW, Park SD, Seo KW. The Index of Microcirculatory Resistance after Primary Percutaneous Coronary Intervention Predicts Long-Term Clinical Outcomes in Patients with ST-Segment Elevation Myocardial Infarction. J Clin Med. 2021 Oct 16;10(20):4752. doi: 10.3390/jcm10204752. PMID 34682875
- [Background] Riley RD, Ensor J, Snell KIE, Harrell FE Jr, Martin GP, Reitsma JB, Moons KGM, Collins G, van Smeden M. Calculating the sample size required for developing a clinical prediction model. BMJ. 2020 Mar 18;368:m441. doi: 10.1136/bmj.m441. No abstract available. PMID 32188600
- [Background] Lewis EF, Moye LA, Rouleau JL, Sacks FM, Arnold JM, Warnica JW, Flaker GC, Braunwald E, Pfeffer MA; CARE Study. Predictors of late development of heart failure in stable survivors of myocardial infarction: the CARE study. J Am Coll Cardiol. 2003 Oct 15;42(8):1446-53. doi: 10.1016/s0735-1097(03)01057-x. PMID 14563590